CLINICAL TRIAL: NCT07117565
Title: Comparison of Intrathecal Dexmedetomidine Versus Intrathecal Fentanyl as Adjuvants to Bupivacaine on Post-Operative Urinary Retention in Lower Limb Surgery
Brief Title: D-FAB-POUR Trial: Dexmedetomidine vs Fentanyl as Adjuvants to Bupivacaine on Postoperative Urinary Retention
Acronym: D-FAB-POUR
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Sujan Dhakal, MD, Principal Investigator, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: D-FAB-POUR Trial
Record Dates: First submitted 2025-06-30; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-06

CONDITIONS: Spinal Anesthesia; Postoperative Complications; Dexmedetomidine; Fentanyl; Anesthesia, Spinal; Bupivacaine; POUR; Orthopedic Surgery; Urinary Retention Postoperative
Keywords: Postoperative urinary retention; Spinal anesthesia; Intrathecal adjuvants; Dexmedetomidine; Fentanyl; Perioperative complications
MeSH Terms: conditions — Postoperative Complications | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: This is a parallel assignment interventional study in which participants are randomly assigned to one of two groups in a 1:1 ratio. One group receives intrathecal dexmedetomidine as an adjuvant to bupivacaine, and the other group receives intrathecal fentanyl with bupivacaine. Each participant receives only one of the study interventions throughout the trial, and no crossover occurs between groups. The study follows a prospective, double-blind, randomized controlled trial design, ensuring both the participants and investigators are blinded to group allocation.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: In this double-blind study, both the participants and the care providers (anesthesiologists) will be blinded to group allocation. The study drugs will be prepared in identical syringes by an independent assistant who is not involved in patient care or outcome assessment. Outcome assessors responsible for measuring postoperative urinary retention and other clinical parameters will also be masked. However, the data analyst will not be blinded to group assignments during statistical analysis, as unblinded data will be required for appropriate group comparisons.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Dexmedetomidine Group (Group BD) (Experimental): Participants in this arm will receive 15 mg (3 mL) of 0.5% hyperbaric bupivacaine combined with 10 mcg (0.5 mL) of dexmedetomidine intrathecally. The total injected volume will be 3.5 mL.
  Interventions: Drug: Intervention 1: Intrathecal Dexmedetomidine with Bupivacaine
- Arm 2: Fentanyl Group (Group BF) (Active Comparator): Participants in this arm will receive 15 mg (3 mL) of 0.5% hyperbaric bupivacaine combined with 25 mcg (0.5 mL) of fentanyl intrathecally. The total injected volume will be 3.5 mL.
  Interventions: Drug: Intervention 2: Intrathecal Fentanyl with Bupivacaine

INTERVENTIONS:
Drug: Intervention 1: Intrathecal Dexmedetomidine with Bupivacaine — Intervention 1: Intrathecal Dexmedetomidine with Bupivacaine
  Detailed Description:
  This intervention consists of a single intrathecal injection of 10 micrograms of dexmedetomidine combined with 15 mg (3 mL) of 0.5% hyperbaric bupivacaine, administered during spinal anaesthesia for lower limb surgery. The total volume administered is 3.5 mL. Dexmedetomidine is an alpha-2 non-opioid adjuvant used as a spinal adjuvant for enhancing analgesia
  Arms: Arm 1: Dexmedetomidine Group (Group BD)
Drug: Intervention 2: Intrathecal Fentanyl with Bupivacaine — This intervention consists of a single intrathecal injection of 25 micrograms of fentanyl combined with 15 mg (3 mL) of 0.5% hyperbaric bupivacaine, administered during spinal anesthesia for lower limb surgery. The total volume administered is 3.5 mL. Fentanyl is a lipophilic opioid commonly used as a spinal adjuvant for enhancing analgesia. This arm is being compared with dexmedetomidine to evaluate differences in POUR incidence, analgesic effectiveness, and side effect profiles.
  Arms: Arm 2: Fentanyl Group (Group BF)

SUMMARY:
This study aims to compare two medications, dexmedetomidine and fentanyl, when used alongside a commonly used spinal anesthetic called bupivacaine in patients undergoing lower limb surgery. The main focus of the study is to see which combination causes fewer problems with urination after surgery - a condition known as postoperative urinary retention (POUR). POUR can lead to discomfort, delayed recovery, and a need for catheterization. Dexmedetomidine is a newer drug that may help reduce this problem compared to fentanyl, which is more commonly used but may increase the risk of urinary retention. This trial will help determine which medication combination provides better pain relief while reducing urinary side effects. The study is being conducted as a randomized, double-blind trial at a hospital in Nepal and will include 190 adult patients.

-

DETAILED DESCRIPTION:
Spinal anaesthesia is a common and effective method used to manage pain during lower limb surgeries. It allows patients to remain awake and comfortable while providing excellent pain control. To make spinal anaesthesia last longer and provide better pain relief, certain medications called adjuvants are added to the main anaesthetic drug, bupivacaine. Two commonly used adjuvants are fentanyl, an opioid, and dexmedetomidine, a medication that works on the body's alpha-2 receptors to provide sedation and pain relief.

However, a known side effect of spinal anaesthesia especially when combined with certain adjuvants is postoperative urinary retention (POUR). This condition occurs when a patient is unable to urinate normally after surgery. POUR can be uncomfortable, may delay recovery, and often requires insertion of a urinary catheter, which can increase the risk of infection and hospital stay.

This clinical trial, called the D-FAB POUR Trial, is designed to find out which of these two adjuvants dexmedetomidine or fentanyl is more likely to cause or prevent POUR when used with bupivacaine in patients undergoing elective lower limb surgery.

The study will involve 190 adult patients. Each participant will receive spinal anaesthesia with bupivacaine and be randomly assigned to also receive either dexmedetomidine or fentanyl. Neither the patients nor the doctors will know which medication is given in a process known as double-blinding to ensure fairness and eliminate bias.

The researchers will monitor the ability of patients to urinate at the third and sixth hours after surgery, using ultrasound to measure bladder volume. If the patient is unable to pass urine and the bladder is overly full, temporary or longer-term catheterisation may be needed. These outcomes will help determine how each drug affects bladder function.

In addition to urinary outcomes, the study will also look at side effects like nausea, vomiting, itching, changes in blood pressure or heart rate, sedation level, and how much extra pain relief the patient needs after surgery.

The goal of this research is to help doctors choose the best adjuvant to use in spinal anaesthesia, one that provides effective pain control without increasing the risk of urinary problems. The findings may lead to improved safety, comfort, and recovery for patients undergoing lower limb operations.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 60 years
* Scheduled for elective lower limb surgery under spinal anesthesia
* Classified as American Society of Anesthesiologists (ASA) physical status II or III
* Minimum height of 150 cm (to ensure uniform drug volume)
* Able to understand the study procedures and provide written informed consent (in English or Nepali)

Exclusion Criteria:

* Contraindications to spinal anesthesia (e.g., coagulopathy, infection at injection site, hemodynamic instability)
* Known allergy or hypersensitivity to bupivacaine, fentanyl, or dexmedetomidine
* Chronic pain conditions or long-term opioid use
* Neurological, Cardiac, Renal, or uncontrolled diabetic conditions
* Current treatment for prostatic pathology or use of alpha-2 blockers
* Presence of a Foley's catheter preoperatively
* Estimated surgical duration: >2.5 hours
* Inability or unwillingness to provide informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 190 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-09-14 (Estimated); Study Completion 2026-11-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Urinary Retention (POUR) at the 3rd Postoperative Hour | 3 hours after spinal anesthesia
  The primary outcome is the number of participants who are unable to void urine at the 3rd postoperative hour with a urinary bladder (UB) volume of ≥600 mL, confirmed by bladder ultrasound. Participants meeting this criterion will be considered to have postoperative urinary retention and will undergo in-out catheterization.

SECONDARY OUTCOMES:
Requirement of Urinary Catheterization at 6th Postoperative Hour | 6 hours after spinal anesthesia
  Number of participants unable to void urine by the 6th postoperative hour, requiring insertion of a Foley's catheter.

CONTACTS AND LOCATIONS:
Locations (1):
- Om Sai Pathibhara Hospital, Bhadrapur, Koshi, Nepal

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to primary and secondary outcomes (including urinary retention, adverse events, and analgesic requirement) will be made available upon reasonable request from qualified researchers. Data will be shared after publication of the main study findings. Access will require a data use agreement and approval by the principal investigator and ethical committee.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 6 months after publication of the primary study results in a peer-reviewed journal.
Access Criteria: Who will have access:
  Qualified researchers, academic collaborators, and clinicians involved in similar fields of study may request access to the de-identified individual participant data (IPD).
  What will be accessible:
  De-identified datasets related to primary and secondary outcomes - including incidence of postoperative urinary retention (POUR), hemodynamic data, sedation scores, rescue analgesic use, and adverse events. Supporting documents such as the study protocol, statistical analysis plan, and case report forms (CRFs) may also be shared upon request.
  How to access:
  Interested researchers must submit a formal written request to the principal investigator (Dr. Sujan Dhakal, szndkl44@gmail.com) explaining the purpose and scope of the intended data use. Requests will be reviewed by the study team and ethics oversight body. Upon approval, access will be granted through a secure data-sharing agreement, ensuring compliance with confidentiality and ethical standards.